CLINICAL TRIAL: NCT03896360
Title: A Randomized Controlled Pilot Study of the Food Order Behavioral Intervention in Prediabetes
Brief Title: Study of the Food Order Behavioral Intervention in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Louis and Rachel Rudin Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1807019463
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-03

CONDITIONS: Pre Diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food order behavioral intervention plus standard care (Experimental): Subjects will receive standard nutrition counseling and additional carbohydrate-last food order behavioral counseling.
  Interventions: Behavioral: Food order behavioral intervention plus standard care
- Standard care (Other): Subjects will receive standard nutrition counseling.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Food order behavioral intervention plus standard care — Subjects in the Food order behavioral intervention plus standard care will receive standard counseling by a registered dietitian and additional carbohydrate last food order behavioral counseling by a member of the research team at baseline and Weeks 4, 8 and 12.
  Arms: Food order behavioral intervention plus standard care
Behavioral: Standard Care — Subjects will receive standard counseling by a registered dietitian at the baseline visit. Standard counseling will be similarly reinforced at weeks 4, 8 and 12.
  Arms: Standard care

SUMMARY:
Investigators have previously shown that eating carbohydrates after protein or vegetables resulted in reduced glucose and insulin excursions over 180 min in patients with T2DM and in individuals with prediabetes as well. This is an open label, randomized controlled pilot study to assess the efficacy of carbohydrate-last food order behavior in reducing the risk of progression to type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
Intensive diet and lifestyle modifications have been shown to reduce the risk of progression to T2DM in several randomized controlled trials. Key components of standard nutritional counseling include reducing calorie intake and glycemic load. Sequential nutrient ingestion is a novel strategy found to attenuate the glycemic effect of a meal. Investigators have previously shown that ingestion of carbohydrates after protein or vegetables results in reduced glucose and insulin excursions over 180 min in patients with T2DM. In addition, investigators also found that levels of the hunger hormone ghrelin were more suppressed at the end of 3 hours after a meal. Furthermore, investigators found that the glycemic effects of food order apply to individuals with prediabetes as well. This study follows previous research on nutrient order and seeks to determine the metabolic effects of this behavioral intervention in the real world. The study will include two randomized groups who are overweight or obese and are diagnosed with prediabetes. The control group will receive standard nutritional counseling at the start of the study and no instructions to change food order behavior. The intervention group will receive regularly scheduled food order counseling over a period of 16 weeks in addition to standard nutritional counseling at baseline. Anthropometric and metabolic parameters, including insulin sensitivity, will be assessed at baseline and at 16 weeks. The primary aim of this study is to determine the proportion of subjects who achieve 15% or greater improvement in 2 hour glucose on OGTT at 16 weeks. If shown to be effective, this data will inform the design of larger study focused on diabetes prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who are 21 years of age or older
* BMI 25-40 kg/m2
* Pre-diabetes defined by an HbA1c of 5.7-6.4%
* Weight stable (< 5% body weight change over preceding 6 months)
* Provide valid informed consent

Exclusion Criteria:

* Previous diagnosis of T2DM or Hb1A1c greater than or equal to 6.5% or fasting glucose > 125mg/dl on screening or 2 hour glucose greater than or equal to 200 mg/dl on OGTT
* Patients who are on any oral/ injectable medications used to treat diabetes including metformin, sulfonylureas, DPP-4 inhibitors, GLP-1 analogs, SGLT2 inhibitors, glitazones and insulin
* Patients on over the counter or approved weight loss medications
* Pregnant or lactating females
* Previous bariatric surgery
* Psychotropic and/or other medications known to significantly impact weight unless on stable dose for 6 months
* eGFR < 45ml/min
* Significant hepatic, cardiac, gastrointestinal, neurologic or other medical illness that would preclude participation in the study
* Untreated hypothyroidism or other endocrine disorders
* Non-English speaking patients
* Any patient deemed unsuitable in the investigator's opinion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving a normal 2-hour glucose (less than 140mg/dl) and/ or greater than or equal to 15% improvement in 2-hour glucose | 16 weeks
  Effect of food order counseling added to standard care on glucose tolerance in individuals with overweight/obesity and prediabetes as measured by the proportion of participants achieving a normal 2-hour glucose (less than 140mg/dl) and/ or greater than or equal to 15% improvement in 2-hour glucose

CONTACTS AND LOCATIONS:
Overall Officials: Alpana P Shukla, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Comprehensive Weight Control Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No